CLINICAL TRIAL: NCT02306616
Title: Improving Care for Cardiovascular Disease in China: A Collaborative Project of AHA and CSC (CCC Project) - Acute Coronary Syndrome
Brief Title: CCC Project- Acute Coronary Syndrome
Status: Completed | Type: Observational
Sponsor: Beijing Institute of Heart, Lung and Blood Vessel Diseases (Other)
Collaborators: American Heart Association (Other); Chinese Society of Cardiology (Other)
Responsible Party: Principal Investigator, Dong ZHAO, Principal Investigator, Beijing Institute of Heart, Lung and Blood Vessel Diseases
Other Study IDs: CCC-ACS-2014
Record Dates: First submitted 2014-11-29; First posted 2014-12-03 (Estimated); Last update posted 2021-01-27 (Actual); Status verified 2021-01

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective

SUMMARY:
To develop and implement quality improvement programs for the treatment of acute coronary syndrome (ACS) in China based on the successful experience of the AHA-Get with the Guidelines program. This program will use data collection, analysis, feedback, and process improvement to extend the use of evidence-based guidelines throughout the healthcare system and improve patient care of acute coronary syndrome.

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients with discharge diagnosis as acute coronary syndrome (including STEMI, NSTEMI and UAP) in 150 tertiary and 100 secondary hospitals.

Exclusion Criteria:

None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with acute coronary syndrome
Sampling Method: Non-Probability Sample
Enrollment: 124363 (Actual)
Dates: Start 2014-11; Primary Completion 2020-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
The overall composite of 11 performance measures for ACS care | Duration of hospital stay, an expected average of 1 week
  Performance measures for ACS care including:
  1. Proportion of patients received aspirin at arrival
  2. Proportion of patients received fibrinolytic therapy within 30 mins (STEMI)
  3. Proportion of patients received primary percutaneous coronary intervention within 90 mins (STEMI)
  4. Proportion of patients received reperfusion therapy (STEMI)
  5. Proportion of patients with aspirin prescribed at discharge
  6. Proportion of patients with clopidogrel or other P2Y12 inhibitors prescribed at discharge
  7. Proportion of patients with beta-blocker prescribed at discharge
  8. Proportion of patients with statin prescribed at discharge
  9. Proportion of patients received evaluation of left ventricular systolic function
  10. Proportion of left ventricular systolic dysfunction patients with ACEI or ARB prescribed at discharge
  11. Proportion of patients received smoking cessation advice/ counseling

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhao, Ph. D, Principal Investigator — Beijing Institute of Heart, Lung and Blood Vessel Diseases
Locations (1):
- Beijing An Zhen Hospital, Beijing, China

REFERENCES:
- [Result] Hao Y, Liu J, Liu J, Smith SC Jr, Huo Y, Fonarow GC, Ma C, Ge J, Taubert KA, Morgan L, Guo Y, Zhang Q, Wang W, Zhao D; CCC-ACS Investigators. Rationale and design of the Improving Care for Cardiovascular Disease in China (CCC) project: A national effort to prompt quality enhancement for acute coronary syndrome. Am Heart J. 2016 Sep;179:107-15. doi: 10.1016/j.ahj.2016.06.005. Epub 2016 Jun 18. PMID 27595685
- [Result] Yang Q, Wang Y, Liu J, Liu J, Hao Y, Smith SC Jr, Huo Y, Fonarow GC, Ma C, Ge J, Taubert KA, Morgan L, Guo Y, Wang W, Zhou Y, Zhao D; CCC-ACS Investigators. Invasive Management Strategies and Antithrombotic Treatments in Patients With Non-ST-Segment-Elevation Acute Coronary Syndrome in China: Findings From the Improving CCC Project (Care for Cardiovascular Disease in China). Circ Cardiovasc Interv. 2017 Jun;10(6):e004750. doi: 10.1161/CIRCINTERVENTIONS.116.004750. PMID 28606999
- [Result] Zhao G, Zhou M, Ma C, Huo Y, Smith SC Jr, Fonarow GC, Ge J, Han Y, Liu J, Hao Y, Liu J, Wang X, Taubert KA, Morgan L, Zhao D, Nie S; CCC-ACS Investigators. In-Hospital Outcomes of Dual Loading Antiplatelet Therapy in Patients 75 Years and Older With Acute Coronary Syndrome Undergoing Percutaneous Coronary Intervention: Findings From the CCC-ACS (Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome) Project. J Am Heart Assoc. 2018 Mar 30;7(7):e008100. doi: 10.1161/JAHA.117.008100. PMID 29602767
- [Result] Zhou M, Liu J, Hao Y, Liu J, Huo Y, Smith SC Jr, Ge J, Ma C, Han Y, Fonarow GC, Taubert KA, Morgan L, Yang N, Xing Y, Zhao D; CCC-ACS Investigators. Prevalence and in-hospital outcomes of diabetes among patients with acute coronary syndrome in China: findings from the Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome Project. Cardiovasc Diabetol. 2018 Nov 27;17(1):147. doi: 10.1186/s12933-018-0793-x. PMID 30482187
- [Result] Xing Y, Liu J, Hao Y, Liu J, Huo Y, Smith SC Jr, Ge J, Ma C, Han Y, Fonarow GC, Taubert KA, Morgan L, Yang N, Zhou M, Zhao D; CCC-ACS Investigators. Prehospital statin use and low-density lipoprotein cholesterol levels at admission in acute coronary syndrome patients with history of myocardial infarction or revascularization: Findings from the Improving Care for Cardiovascular Disease in China (CCC) project. Am Heart J. 2019 Jun;212:120-128. doi: 10.1016/j.ahj.2019.02.019. Epub 2019 Mar 13. PMID 30986750
- [Result] Yang N, Liu J, Liu J, Hao Y, Huo Y, Smith SC Jr, Ge J, Ma C, Han Y, Fonarow GC, Taubert KA, Morgan L, Zhou M, Xing Y, Zhao D; CCC-ACS Investigators. Performance on management strategies with Class I Recommendation and A Level of Evidence among hospitalized patients with non-ST-segment elevation acute coronary syndrome in China: Findings from the Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome (CCC-ACS) project. Am Heart J. 2019 Jun;212:80-90. doi: 10.1016/j.ahj.2019.02.012. Epub 2019 Mar 4. PMID 30981036
- [Result] Hao Y, Liu J, Liu J, Yang N, Smith SC Jr, Huo Y, Fonarow GC, Ge J, Taubert KA, Morgan L, Zhou M, Xing Y, Ma CS, Han Y, Zhao D. Sex Differences in In-Hospital Management and Outcomes of Patients With Acute Coronary Syndrome. Circulation. 2019 Apr 9;139(15):1776-1785. doi: 10.1161/CIRCULATIONAHA.118.037655. PMID 30667281
- [Derived] Liu Y, Liu X, Sun D, Gu R, Li M, Wang X. Aspirin Combined With Ticagrelor or Clopidogrel in STEMI Patients With Diabetes Mellitus and Poor Glycemic Control Undergoing Primary PCI: A Multicenter Retrospective Cohort Study. Catheter Cardiovasc Interv. 2026 Feb 8. doi: 10.1002/ccd.70503. Online ahead of print. PMID 41656976
- [Derived] Zhou Z, Xie H, Fan F, Yang F, Jiang J, Zheng B, Zhang Y, Hao Y, Liu J, Gong Y, Zhao D, Smith SC, Huo Y. Comparison of in-hospital net clinical outcomes of ticagrelor and clopidogrel in acute coronary syndrome patients stratified by CRUSADE score: findings from the CCC-ACS registry. Platelets. 2025 Dec;36(1):2570743. doi: 10.1080/09537104.2025.2570743. Epub 2025 Oct 27. PMID 41143351
- [Derived] Zhou C, Zhang M, Zhao Z, Li E, Zhao Y, Luo W, Zheng K, Liu Y, Yin C, Zhang X, Gao H, Zhao D, Ma C. Clopidogrel vs. ticagrelor in ST-elevation myocardial infarction complicated by cardiogenic shock undergoing primary PCI : Findings from a National, multicenter registry. Thromb J. 2025 Apr 22;23(1):38. doi: 10.1186/s12959-025-00721-z. PMID 40264117
- [Derived] Zhou C, Zhang M, Zhao Z, Li E, Zhao Y, Wang H, Luo W, Zheng K, Liu Y, Yin C, Zhang X, Gao H, Hou X, Zhao D, Ma C. Safety and efficacy of post-procedure anticoagulation in ST-elevation myocardial infarction complicated by cardiogenic shock undergoing primary percutaneous coronary intervention. BMC Cardiovasc Disord. 2025 Mar 28;25(1):231. doi: 10.1186/s12872-025-04639-2. PMID 40155819
- [Derived] Zhang Y, Hao Y, Liu J, Yang N, Smith SC Jr, Huo Y, Fonarow GC, Ge J, Morgan L, Sun Z, Hu D, Yang Y, Ma CS, Zhao D, Han Y, Liu J, Zeng Y; CCC-ACS Investigators. Percutaneous coronary intervention in patients with acute coronary syndromes and increased platelet count. Arch Cardiovasc Dis. 2025 May;118(5):304-311. doi: 10.1016/j.acvd.2025.01.005. Epub 2025 Feb 13. PMID 39984408
- [Derived] Zhao T, Wang J, Gu R, Sun D, Zheng L, Tian X, Han Y, Wang X; CCC-ACS investigators. Comparison of Multivessel Versus Culprit-Vessel-Only Revascularization in Patients With STEMI and Multivessel Disease During Primary PCI: In-Hospital Outcomes From the CCC-ACS Project in China. Catheter Cardiovasc Interv. 2025 Jan;105(1):43-53. doi: 10.1002/ccd.31332. Epub 2024 Dec 10. PMID 39659090
- [Derived] Yang N, Zhao W, Hao Y, Liu J, Liu J, Zhao X, Yan Y, Nie S, Gong W; CCC investigators. Incidence and risk factors for cardiac rupture after ST-segment elevation myocardial infarction in contemporary era: findings from the improving care for cardiovascular disease in China-Acute Coronary Syndrome project. Intern Emerg Med. 2025 Jan;20(1):77-85. doi: 10.1007/s11739-024-03746-w. Epub 2024 Oct 27. PMID 39463195
- [Derived] Gong W, Yan Y, Liu J, Wang X, Zheng W, Que B, Ai H, Smith SC Jr, Fonarow GC, Morgan L, Zhao D, Ma C, Han Y, Nie S; CCC-ACS Investigators. In-Hospital Mortality and Treatment in Patients With Acute Coronary Syndrome With and Without Standard Modifiable Cardiovascular Risk Factors: Findings From the CCC-ACS Project. J Am Heart Assoc. 2024 Oct;13(19):e029252. doi: 10.1161/JAHA.122.029252. Epub 2024 Sep 18. PMID 39291502
- [Derived] Zhang T, Wang X, Zhang Y, Feng T, Zhou Y, Zhao L. Early beta-blocker use and in-hospital outcomes in patients with chronic obstructive pulmonary disease hospitalized with acute coronary syndrome: findings from the CCC-ACS project. Front Cardiovasc Med. 2024 Jul 11;11:1385943. doi: 10.3389/fcvm.2024.1385943. eCollection 2024. PMID 39055663
- [Derived] Zhao G, Zhou M, Zhao X, Ma C, Han Y, Liu J, Zhao D, Nie S; CCC-ACS Investigators. Characteristics, Treatment, and In-Hospital Outcomes of Older Patients With STEMI Without Standard Modifiable Risk Factors. JACC Asia. 2023 Nov 21;4(1):73-83. doi: 10.1016/j.jacasi.2023.09.013. eCollection 2024 Jan. PMID 38222256
- [Derived] Zhu J, Liu W, Li J, Ma C, Zhao D. A Small Increase in Serum Creatinine within 48 h of Hospital Admission Is an Independent Predictor of In-Hospital Adverse Outcomes in Patients with ST-Segment Elevation Myocardial Infarction Undergoing Primary Percutaneous Coronary Intervention: Findings from the Improving Care for Cardiovascular Disease in the China Project. Cardiol Res Pract. 2023 Mar 28;2023:1374206. doi: 10.1155/2023/1374206. eCollection 2023. PMID 37025394
- [Derived] Wang Y, Geng Y, Zhang O, Xu Q, Xue Y, Zhou B, Zhang P; CCC-ACS Investigators. Association between P2Y12 inhibitor reloading and in-hospital outcomes for patients with non-ST-segment elevation acute coronary syndrome already on chronic P2Y12 receptor inhibitors therapy in China: findings from the CCC-ACS (improving care for cardiovascular disease in China-acute coronary syndrome) project. Eur J Med Res. 2023 Feb 2;28(1):59. doi: 10.1186/s40001-023-01025-6. PMID 36732830
- [Derived] Li Z, Sun H, Hao Y, Liu H, Jin Z, Li L, Zhang C, Ma M, Teng T, Chen X, Shen Y, Yu Y, Liu J, Richards AM, Tan HC, Zhao D, Zhou X, Yang Q. Renin-angiotensin system inhibition and in-hospital mortality in acute coronary syndrome patients with advanced renal dysfunction: findings from CCC-ACS project and a nationwide electronic health record-based cohort in China. Eur Heart J Qual Care Clin Outcomes. 2023 Dec 22;9(8):785-795. doi: 10.1093/ehjqcco/qcad006. PMID 36731865
- [Derived] Yang Y, Hao Y, Liu J, Yang N, Hu D, Sun Z, Zhao D, Liu J; Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome (CCC-ACS) Investigators. Practice of reperfusion in patients with ST-segment elevation myocardial infarction in China: findings from the Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome project. Chin Med J (Engl). 2022 Dec 5;135(23):2821-2828. doi: 10.1097/CM9.0000000000002257. PMID 36728532
- [Derived] Yang N, Liu J, Liu J, Hao Y, Smith JSC, Huo Y, Fonarow GC, Ge J, Morgan L, Ma C, Han Y, Zhao D; Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome (CCC-ACS) project investigators. In-hospital outcomes of ticagrelor versus clopidogrel in patients 75 years or older with acute coronary syndrome: findings from the Improving Care for Cardiovascular Disease in China (CCC)-Acute Coronary Syndrome Project. Age Ageing. 2022 Nov 1;51(11):afac231. doi: 10.1093/ageing/afac231. PMID 36413586
- [Derived] Gong W, Yan Y, Wang X, Zheng W, Smith SC Jr, Fonarow GC, Morgan L, Liu J, Zhao D, Ma C, Han Y, Montalescot G, Nie S; CCC-ACS Investigators. Risk Factors for In-Hospital Cardiac Arrest in Patients With ST-Segment Elevation Myocardial Infarction. J Am Coll Cardiol. 2022 Nov 8;80(19):1788-1798. doi: 10.1016/j.jacc.2022.08.797. PMID 36328690
- [Derived] Wang Y, Yang N, Suo M, Liu X, Wang Z, Zhang X, Liu J, Zhao D, Wu X; CCC-ACS Investigators. In-hospital outcomes of Ticagrelor versus Clopidogrel in high bleeding risk patients with acute coronary syndrome: Findings from the CCC-ACS project. Thromb Res. 2022 Aug;216:43-51. doi: 10.1016/j.thromres.2022.04.004. Epub 2022 May 10. PMID 35714445
- [Derived] Xu S, Li Z, Yang T, Li L, Song X, Hao Y, Smith SC, Fonarow GC, Morgan L, Liu J, Liu J, Zhao D, Yang Q, Zhou X, Li Y. Association between Early Oral beta-Blocker Therapy and Risk for In-Hospital Major Bleeding after Percutaneous Coronary Intervention for Acute Coronary Syndrome: Findings from CCC-ACS Project. Eur Heart J Qual Care Clin Outcomes. 2022 Jun 17:qcac036. doi: 10.1093/ehjqcco/qcac036. Online ahead of print. PMID 35713509
- [Derived] Lin YW, Huang JL, Wei XB, Jiang M, Ran P, Li J, Qiu J, Zhong Q, Zhou YL, Chen JY, Yu DQ. Estimated glomerular filtration rate derived from different formulas and prognosis in acute coronary syndrome: Findings from the improving care for cardiovascular disease in China-acute coronary syndrome project. Am J Med Sci. 2022 Nov;364(5):565-574. doi: 10.1016/j.amjms.2021.10.034. Epub 2022 Jun 2. PMID 35660542
- [Derived] Yang JQ, Ran P, Li J, Zhong Q, Smith SC Jr, Wang Y, Fonarow GC, Qiu J, Morgan L, Wei XB, Chen XB, Huang JL, Hao YC, Zhou YL, Siu CW, Zhao D, Chen JY, Yu DQ. A Risk Stratification Scheme for In-Hospital Cardiogenic Shock in Patients With Acute Myocardial Infarction. Front Cardiovasc Med. 2022 Mar 4;9:793497. doi: 10.3389/fcvm.2022.793497. eCollection 2022. PMID 35310985
- [Derived] Zhou M, Zhang J, Liu J, Smith SC Jr, Ma C, Ge J, Huo Y, Fonarow GC, Liu J, Hao Y, Gao F, Sun Y, Morgan L, Yang N, Hu G, Zeng Y, Han Y, Zhao D; CCC-ACS Investigators. Proton Pump Inhibitors and In-Hospital Gastrointestinal Bleeding in Patients With Acute Coronary Syndrome Receiving Dual Antiplatelet Therapy. Mayo Clin Proc. 2022 Apr;97(4):682-692. doi: 10.1016/j.mayocp.2021.11.037. Epub 2022 Feb 12. PMID 35164933
- [Derived] Wang X, Zhao G, Zhou M, Ma C, Ge J, Huo Y, Smith SC Jr, Fonarow GC, Hao Y, Liu J, Morgan L, Gong W, Yan Y, Liu J, Zhao D, Han Y, Nie S. Trends in Bleeding Events Among Patients With Acute Coronary Syndrome in China, 2015 to 2019: Insights From the CCC-ACS Project. Front Cardiovasc Med. 2021 Dec 13;8:769165. doi: 10.3389/fcvm.2021.769165. eCollection 2021. PMID 34966795
- [Derived] Yang Q, Sun D, Pei C, Zeng Y, Wang Z, Li Z, Hao Y, Song X, Li Y, Liu G, Tang Y, Smith SC, Han Y, Huo Y, Ge J, Ma C, Fonarow GC, Morgan L, Liu J, Liu J, Zhou M, Zhao D, Zhou Y, Zhou X; CCC-ACS Investigators. LDL cholesterol levels and in-hospital bleeding in patients on high-intensity antithrombotic therapy: findings from the CCC-ACS project. Eur Heart J. 2021 Aug 31;42(33):3175-3186. doi: 10.1093/eurheartj/ehab418. PMID 34347859
- [Derived] Yang L, Ye N, Wang G, Bian W, Xu F, Zhao D, Liu J, Hao Y, Liu J, Yang N, Cheng H; CCC-ACS. The association between atrial fibrillation and in-hospital outcomes in chronic kidney disease patients with acute coronary syndrome: findings from the improving care for cardiovascular disease in China-acute coronary syndrome (CCC-ACS) project. BMC Cardiovasc Disord. 2021 Jul 17;21(1):345. doi: 10.1186/s12872-021-02125-z. PMID 34273963
- [Derived] Ran P, Yang JQ, Li J, Li G, Wang Y, Qiu J, Zhong Q, Wang Y, Wei XB, Huang JL, Siu CW, Zhou YL, Zhao D, Yu DQ, Chen JY. A risk score to predict in-hospital mortality in patients with acute coronary syndrome at early medical contact: results from the Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome (CCC-ACS) Project. Ann Transl Med. 2021 Jan;9(2):167. doi: 10.21037/atm-21-31. PMID 33569469
- [Derived] Zhao X, Kang Y, Wang X, Yang X, Ai G, Liu Y, Xu P, Zhang J, Gu C, Zhang Y, Hao Y, Zhao D, Han Y; CCC investigators. Clinical significance of glycated hemoglobin in acute coronary syndrome patients from the CCC-ACS project : Findings from a multicenter retrospective observational study. Herz. 2021 Sep;46(Suppl 2):287-294. doi: 10.1007/s00059-020-04999-9. Epub 2020 Nov 24. PMID 33231709
- [Derived] Hu G, Zhou M, Liu J, Smith SC Jr, Ma C, Ge J, Huo Y, Fonarow GC, Hao Y, Liu J, Taubert KA, Morgan L, Yang N, Zeng Y, Han Y, Zhao D; CCC-ACS Investigators. Smoking and Provision of Smoking Cessation Interventions among Inpatients with Acute Coronary Syndrome in China: Findings from the Improving Care for Cardiovascular Disease in China-Acute Coronary Syndrome Project. Glob Heart. 2020 Oct 23;15(1):72. doi: 10.5334/gh.784. PMID 33150137
- [Derived] Ye N, Yang L, Wang G, Bian W, Xu F, Ma C, Zhao D, Liu J, Hao Y, Liu J, Yang N, Cheng H; CCC-ACS. Admission fasting plasma glucose is associated with in-hospital outcomes in patients with acute coronary syndrome and diabetes: findings from the improving Care for Cardiovascular Disease in China - Acute Coronary Syndrome (CCC-ACS) project. BMC Cardiovasc Disord. 2020 Aug 20;20(1):380. doi: 10.1186/s12872-020-01662-3. PMID 32819275